CLINICAL TRIAL: NCT05102526
Title: The Impact of a School-based Program on the Psychological Health of Young Adolescents: The Facilitator Role of a Teacher Component and Content Delivered in the School
Brief Title: Increasing the Impact of a School Prevention Program Among Young Adolescents by Adding a Teacher Component
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tel-Hai
Record Dates: First submitted 2021-10-23; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Primary Prevention
Keywords: prevention-program; Physical assessment; self-esteem; self-care; Teachers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Young Millie" prevention program, active teachers (Experimental): The "Young Mili" program will be delivered to teens ages 10-12, over 3 months. The program contains nine 90-minute weekly sessions focusing on media literacy, self-esteem, self-esteem and physical self-esteem. Teachers will also participate by delivering planned activities to their students in addition to each week's theme, in parallel with an externally delivered program. All participants will complete a self-report questionnaire at the beginning of the study, after the end of the program and three months after the end of the program.
  Interventions: Behavioral: Experimental: "Young Millie" prevention program, active teachers
- "Young Mili" prevention program, passive teachers (Active Comparator): The "Young Mili" program will be delivered to teens ages 10-12, over 3 months. The program contains nine 90-minute weekly sessions focusing on media literacy, self-esteem, self-esteem and body image. Teachers will not participate in the program, they will be present in class only during the program on transfer abroad. All participants will complete a self-report questionnaire at the beginning of the study, after the end of the program and three months after the end of the program.
  Interventions: Behavioral: Prevention program: "Young Mili", non active teachers

INTERVENTIONS:
Behavioral: Experimental: "Young Millie" prevention program, active teachers — Prevention program: "Young Mili", in collaboration with the teacher
  Arms: "Young Millie" prevention program, active teachers
Behavioral: Prevention program: "Young Mili", non active teachers — Prevention program: "Young Mili", without the participation of the teacher
  Arms: "Young Mili" prevention program, passive teachers

SUMMARY:
A randomized clinical trial in clusters, including the development and implementation of an intervention program among young adolescents and their teachers. The research hypothesis is that the intervention program will yield improvement in adolescents whose parents participated in the program, compared with adolescents whose teachers were not involved in the intervention. The results will be measured using the research questionnaire, which participants will complete before, after and three months after the end of the program. The questionnaire will include approved questionnaires with good psychometric properties. In addition, there will be a quality interview. The study protocol was approved by the Tel Hai College Institutional Audit Committee. Parents of all participants in the intervention and control group as well as the teachers involved in the program received information about the program and research and were asked to give informed consent.

DETAILED DESCRIPTION:
Early adolescence (10-13 years) is characterized by hormonal changes and accelerated physiological growth. Significant risk factors for the physical and mental health of children and adolescents include, among other things, reduced physical activity, low self-esteem and self-esteem.

"Mili - a unique shield for daily resilience" is a preventive intervention program. The main goal of the program is to increase the self-care behaviors and self esteem of adolescents and prevent negative physical self-image, as well as to develop media literacy. In this study, researchers will focus on a school-based program designed for ages 10-12, grades 5-6, with a primary goal to develop self-care, media literacy, self-esteem, and positive body image. To increase the impact of the "Young Mili" program on adolescents, the researchers developed a teacher component as an adjunct to the school-based intervention, usually facilitated only by college students. The study will first evaluate the impact of teachers on the program, and then evaluate the difference between adolescent outcomes from the program with or without this supplement.

The results will be measured using the research questionnaire, to be completed by the participants (both teachers and adolescents) before, after, and three months after the end of the program. The questionnaire will include validated scales with good psychometric properties. In addition, qualitative interviews will be conducted among teachers. The study protocol was approved by the Tel Hai College Institutional Audit Committee. Parents of all participants, in the intervention and the control group, as well as teachers involved in the program, were given information about the program and the research and were asked to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Teachers of elementary school classes
* 10-12-year-old students of participating teachers
* Participants who filled out the questionnaires before and after the program
* Participants whose parents signed a letter of informed consent.

Exclusion Criteria:

* Participants who didn't complete the questionnaires at baseline or at least twice.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Sociocultural Attitudes towards Appearance Questionnaire-4, Affects by Media subscale. | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  The Sociocultural Attitudes Towards Appearance Questionnaire (Schaefer et al., 2015). The investigators included the Media subscale, including 4 items. Items are rated on a 5-point scale: (1) always, (2) often, (3) sometimes, (4) rarely, (5) never. The total score is based on computing the average. A higher score indicates higher pressure from the media to change one's look.
Change from Baseline in Rosenberg Self Esteem Scale | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  Rosenberg Self Esteem Scale (Rosenberg, 1965)- 10 items. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or "strongly disagree" on items 1, 3, 4, 7, 10, and "strongly agree" or "agree" on items 2, 5, 6, 8, 9. Two or three out of three correct responses to items 3, 7, and 9 are scored as one item. One or two out of two correct responses for items 4 and 5 are considered as a single item; items 1,8, and 10 are scored as individual items; and combined correct responses (one or two out of two) to items 2 and 6 are considered to be a single item.
Change from Baseline in Body Esteem Scale | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  Body Esteem Scale- This questionnaire examines self-esteem of body and physical appearance and consists of 3 subscales: appearance (10 items), weight (8 items) and attribution 187 to others (5 items). Items are rated on a 5-point scale: (1) never, (2) rarely, (3) sometimes, (4) 188 often, and (5) always. A higher score indicates higher body-esteem (Mendelson, Mendelson, & White, 2001)
Change from Baseline in Advertising Scale | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  The Advertising scale contains 1 item- Identification of strategies used by media. This question is reflected as a protective factor. It contains 8 different strategies which participants choose from: higher number of strategies identified indicate better media literacy. (Golan et al., 2013).
Change from Baseline in Self-Care behaviors | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  Developed by Prof. Moria Golan and assessed in previous research. Includes 14 items which are rated on a 4-point scale: (1) never, (2) rarely, (3) sometimes, (4) always. Items are summed, and higher scores indicate higher self-care behaviors. This questionnaire was designed to assess self care behaviors in adolescents.

SECONDARY OUTCOMES:
Change from Baseline in The Connor-Davidson Resilience Scale (CD-RISC) | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the course, measuring a change in scores
  The CD-RISC is based on Connor and Davidson's operational definition of resilience, which is the ability to "thrive in the face of adversity." The scale includes 25 items, from 5 sub-scales:

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Hai College, Kiryat Shmona, Upper Galilee, Israel

IPD SHARING:
Plan to Share IPD: Undecided